CLINICAL TRIAL: NCT07239661
Title: The Clinical Efficacy of Electroacupuncture Combined With PD-1 Inhibitor in the Treatment of ECOG2 Advanced Non-small Cell Lung Cancer
Brief Title: Electroacupuncture Combined With PD-1 Inhibitor for ECOG2 Advanced NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kong Fanming (Other)
Responsible Party: Sponsor-Investigator, Kong Fanming, Director of Oncology Department, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Organization: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TYLL2025[K]016
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer; Electroacupuncture; PD-1 Inhibitors; ECOG PS 2 Points
Keywords: electroacupuncture; Immunotherapy; immune checkpoint inhibitor; Non-Small Cell Lung Cancer; ECOG PS 2 points
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Due to the specific nature of acupuncture clinical research, it is challenging to achieve double blinding of subjects and operators. Therefore, this trial was blinded to subjects and statisticians only. The statistical analyst was a non-subject and was not aware of the patient's treatment or the trial protocol. For all patients who participated in acupuncture, blinded evaluation questions were asked one week after acupuncture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EA + ICIs group (Experimental): Bilateral Zusanli (ST36) and Sanyinjiao (SP6) acupoints were selected. After obtaining deqi sensation upon needle insertion, an electroacupuncture device was connected to each of the selected acupoints. A sparse-dense wave mode was chosen, with an intensity ranging from 0.5 to 2 mA, adjusted according to patient tolerance. The needles were retained for 20 minutes before removal. The electroacupuncture treatment was initiated on the same day as the commencement of the immunotherapy cycle, administered once daily for a total of five sessions, ensuring that each immunotherapy cycle was synchronized with electroacupuncture treatment. The overall treatment consisted of 4 to 6 cycles.
  Interventions: Other: Electroacupuncture (EA)
- Sham EA + ICIs group (Sham Comparator): Bilateral Zusanli (ST36) and Sanyinjiao (SP6) acupoints were selected. Electroacupuncture devices were connected to these acupoints. A sparse-dense wave mode was utilized, with an intensity ranging from 0.5 to 2 mA, and the needles were retained for 20 minutes before removal. In the sham electroacupuncture group, no manual manipulation was performed. The placement of electrodes and other treatment settings were identical to those in the electroacupuncture group, but without skin penetration, electrical output, or needling techniques to induce deqi. Electroacupuncture treatment was initiated on the same day as the start of the immunotherapy cycle, administered once daily for a total of five sessions, ensuring synchronization with each immunotherapy cycle. The overall treatment regimen consisted of 4 to 6 cycles.
  Interventions: Other: Sham electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture (EA) — In the electroacupuncture group, bilateral Zusanli (ST36) and Sanyinjiao (SP6) points were selected for needling. Upon achieving the "deqi" sensation, the electroacupuncture device was connected to the needles at both points. A dispersed-dense wave was applied with an intensity ranging from 0.5 to 2 mA, adjusted according to the patient's tolerance. The needles were retained for 20 minutes, after which they were removed.
  Arms: EA + ICIs group
Other: Sham electroacupuncture — In the sham electroacupuncture group, bilateral Zusanli (ST36) and Sanyinjiao (SP6) points were selected for sham electroacupuncture intervention, which did not receive manual manipulation. The electrode placement and other treatment settings were identical to those in the electroacupuncture group, but no skin penetration, electrical output, or needle techniques were applied to induce the sensation of "deqi." No genuine electroacupuncture stimulation was administered in this group.
  Arms: Sham EA + ICIs group

SUMMARY:
The aim of this study was to systematically evaluate the clinical efficacy and safety of electroacupuncture (EA) combined with PD-1 inhibitors in patients with advanced non-small cell lung cancer (NSCLC) who have an ECOG performance status of 2 through a multicenter, randomized, sham-controlled clinical trial. The core scientific question addressed in this study was whether EA combined with standard immunotherapy could further improve progression-free survival (PFS), immune function, and quality of life in these patients. Patients meeting the inclusion criteria were randomly assigned in a 1:1 ratio to receive EA plus a PD-1 inhibitor (trial group) or sham EA plus a PD-1 inhibitor (control group) through a computerized randomization system. PD-1 inhibitors were administered every 21 days for four to six cycles, followed by maintenance therapy according to each patient's condition. EA intervention was initiated on the first day of each immunotherapy cycle and administered once daily for five sessions per cycle, continuing for four to six cycles. The primary endpoint was progression-free survival (PFS). The secondary endpoints included objective response rate (ORR), overall survival (OS), first-line treatment completion rate, quality of life as assessed by the EORTC QLQ-C30 scale, traditional Chinese medicine (TCM) syndrome score, immune function index, and incidence of adverse events according to CTCAE 5.0 criteria. In addition, peripheral blood was collected from patients at baseline for non-coding RNA sequencing, and differentially expressed genes were identified through bioinformatics analysis to determine potential molecular biomarkers associated with the synergistic effects of EA, thereby providing a basis for accurately identifying patients likely to benefit from EA therapy.

DETAILED DESCRIPTION:
Based on the principles of evidence-based medicine, a randomized controlled clinical trial was conducted to provide high-quality evidence on the clinical efficacy and immunomodulatory effects of acupuncture combined with first-line immunotherapy in patients with advanced NSCLC with an ECOG PS2, thereby facilitating the promotion and application of "precision" traditional Chinese medicine (TCM) treatment. This project provides an evidence-based reference for developing standardized treatment protocols and clinical pathways for advanced NSCLC and further clarifies the potential role of TCM within the therapeutic framework of advanced lung cancer, holding significant academic value and substantial social benefits.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage ⅢB-Ⅳ non-small cell lung cancer (NSCLC) confirmed by pathological or cytological examination;
* Patients with negative driver gene mutations, excluding those harboring EGFR mutations, ALK rearrangements, or other common driver gene alterations as determined by genetic testing or other molecular biological methods;
* An Eastern Cooperative Oncology Group (ECOG) performance status score of 2;
* A programmed death-ligand 1 (PD-L1) tumor proportion score (TPS) ≥ 1%;
* An expected survival time of more than 3 months, as assessed by the clinician based on the patient's overall condition, tumor progression, and response to treatment;
* Patients with good treatment compliance who provided written informed consent, confirming their understanding of and willingness to undergo treatment and follow-up according to the study protocol.

Exclusion Criteria:

* Patients with a history or concurrent diagnosis of other malignant tumors within the past five years;
* Patients with severe organ impairment or serious comorbidities, such as cardiac dysfunction (New York Heart Association [NYHA] class Ⅲ-Ⅳ), hepatic or renal insufficiency, as determined by standard clinical examinations including liver and kidney function tests and electrocardiography;
* Patients with untreated central nervous system (CNS) metastases were excluded; eligible patients were required to have stable disease confirmed by imaging after receiving at least one systemic or surgical treatment;
* Patients with psychiatric disorders, including schizophrenia or bipolar disorder, particularly those requiring pharmacologic treatment;
* Patients with a history of multiple drug allergies, an allergic predisposition, or a history of severe allergic reactions such as anaphylactic shock or allergic rash;
* Subjects with active autoimmune or infectious diseases, including but not limited to chronic viral hepatitis, active pulmonary tuberculosis, or other infections or autoimmune disorders deemed by clinicians to potentially affect the study;
* Female patients who were pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | Defined as the time interval from the date of enrollment to the first documented occurrence of disease progression or death from any cause, whichever comes first. This outcome will be assessed up to 100 months.
  Defined as the interval from the time of enrollment to the first documentation of disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
This decision may stem from concerns regarding privacy or ethical issues associated with data sharing, or because the research data is considered proprietary and not intended for public disclosure.